CLINICAL TRIAL: NCT04243668
Title: ENDOSCOPIC ANTI REFLUX MUCOSAL ABLATION THERAPHY (ARMA) FOR THE TREATMENT OF PROTON PUMP INHIBITOR DEPENDENT GASTRO ESOPHAGEALREFLUX DISEASE: OPEN LABEL SINGLE CENTER OBSERVATIONAL STUDY
Brief Title: ANTI REFLUX MUCOSAL ABLATION THERAPHY (ARMA)
Acronym: ARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, PRINCIPAL INVESTIGATOR, Asian Institute of Gastroenterology, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARMA01
Record Dates: First submitted 2020-01-07; First posted 2020-01-28 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANTI REFLUX MUCOSAL ABLATION THERAPHY (Experimental): In patients fulfilling inclusion criteria and willing for ARMA, the procedure involves ablation of the mucosa of the EGJ using TT knife (ARMA). Subsequently, saline solution mixed with indigo-carmine is injected at the submucosa level to raise a submucosal bleb, followed by ablation of the mucosa along the lesser curvature using TT knife.The approximate duration of the procedure is 40min.
  Interventions: Procedure: ANTI REFLUX MUCOSAL ABLATION THERAPHY (ARMA)

INTERVENTIONS:
Procedure: ANTI REFLUX MUCOSAL ABLATION THERAPHY (ARMA) — In patients fulfilling inclusion criteria and willing for ARMA, the procedure involves ablation of the mucosa of the EGJ using TT knife (ARMA). Subsequently, saline solution mixed with indigo-carmine is injected at the submucosa level to raise a submucosal bleb, followed by ablation of the mucosa along the lesser curvature using TT knife.The approximate duration of the procedure is 40min.
  Follow up will include objective evaluation of reflux disease with: upper endoscopy, esophageal manometry, pHmetry,reflux questionnaire.

SUMMARY:
OBJECTIVES To study the safety and efficacy of Endoscopic Anti Reflux Mucosal Ablation (ARMA) procedure for the treatment of proton pump inhibitor (PPI) dependent gastro-esophageal reflux disease (GERD)

DESIGN OF THE Prospective interventional study Sample size: 216

DETAILED DESCRIPTION:
In patients fulfilling inclusion criteria and willing for ARMA, the procedure involves ablation of the mucosa of the EGJ using TT knife (ARMA). Subsequently, saline solution mixed with indigo-carmine is injected at the submucosa level to raise a submucosal bleb, followed by ablation of the mucosa along the lesser curvature using TT knife.The approximate duration of the procedure is 40min.

Submucosal injection and elevation will not be used as a part of ARMA procedure for 10 patients amended protocol version 2.0

Follow up will include objective evaluation of reflux disease with: upper endoscopy, esophageal manometry, pHmetry,reflux questionnaire.

Inclusion criteria

* Patients (between 18 to 60 years of age) with PPI dependent GERD and pathologic esophageal acid exposure as documented by percentage time esophageal PH less than 4 of more than 4.2% on PH-metry during 24-hrs period while off PPI
* Patients who are willing to pay the expenses of the ARMA procedure

Exclusion criteria

* Large Hiatal hernia >3cm
* Gr C/D esophagitis
* Lower esophageal sphincter (LES) pressure<5 or >15 mm Hg
* Paraesophageal hernia
* GE flap valve grade IV (Hill's classification)
* Barretts esophagus
* Esophageal dysmotility
* ASA physical status >II
* Previous esophageal or gastric surgery
* Pregnancy

Patients screening and inclusion:

The study will be conducted over 6-months period. Data of patients presenting with PPI dependent GERD will be recorded and maintained. At initial screening, GERD HRQL and requirement of anti-secretory medicines (detailed drug history) will be assessed along with gastroscopy. All anti-secretory medicines will be stopped for 7 days and GERD HRQL will be reassessed off drugs. Esophageal high resolution manometry with 24-h pH impedance monitoring will be done on the 8th day after stopping medicines. Basal LES pressure, esophageal motility pattern, 24-h esophageal acid exposure, non acidic bolus reflux, number of reflux episodes, DeMeester score, symptom index and symptom association probability would be assessed.Those patients with pathologic esophageal acid exposure as described previously will be included in the trial. Patients will then be directly assigned by a computer to ARMA procedure. The principle investigator and the study coordinators would be open label to the treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients (between 18 to 60 years of age) with PPI dependent GERD and pathologic esophageal acid exposure as documented by percentage time esophageal PH less than 4 of more than 4.2% on PH-metry during 24-hrs period while off PPI

  * Patients who are willing to pay the expenses of the ARMA procedure

Exclusion Criteria:

* • Large Hiatal hernia >3cm

  * Gr C/D esophagitis
  * Lower esophageal sphincter (LES) pressure<5 or >15 mm Hg
  * Paraesophageal hernia
  * GE flap valve grade IV (Hill's classification)
  * Barretts esophagus
  * Esophageal dysmotility
  * ASA physical status >II
  * Previous esophageal or gastric surgery
  * Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Gastro esophageal reflux disease symptoms by more than 50% from baseline at 3 months | 3 months
  Improvement in Gastroesophageal reflux disease symptoms by more than 50% from baseline at 3 months which would be assessed based on visual analog scale VAS 0 LOW SCORE 10 WORSE SYMPTOM SCORE

SECONDARY OUTCOMES:
requirement of PPI at 3, 6 and 12 months | requirement of PPI at 3, 6 and 12 months
  requirement of Proton Pump Inhibitors at 3, 6 and 12 months based on GERD score evaluated based on visual analog scale VAS 0 LOW SCORE 10 WORSE SYMPTOM SCORE
Improvement in esophageal acid exposure | 6 months
  Improvement in esophageal acid exposure in PH impedence monitoring report from baseline
Improvement in lower esophageal sphincter pressure at 3 months | 12 months
  Improvement in lower esophageal sphincter pressure at 3 months i.e sphincter pressure will be less compare to baseline pressure which will be known by the Esophageal manometry report.

CONTACTS AND LOCATIONS:
Overall Officials: Nageshwar Reddy, DNB, Principal Investigator — Chairman
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koduri KK, Singla N, Maragoni RG, Jagtap N, Singh AP, Kalapala R, Reddy DN. Efficacy and safety of anti-reflux mucosal ablation therapy at 12 months. Indian J Gastroenterol. 2025 Oct;44(5):700-707. doi: 10.1007/s12664-025-01761-z. Epub 2025 Jun 11. PMID 40498286